CLINICAL TRIAL: NCT04428606
Title: Placebo Controlled Pilot Trial to Determine the Effect of Metabolic Rheostat™ and Butyrate Ultra on Hemoglobin A1C and Blood Glucose Levels in Patients With Pre-diabetes
Brief Title: Study to Determine the Effect of Synbiotics in Patients With Pre-diabetes
Acronym: Rheostat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhaoping Li (Other)
Responsible Party: Sponsor-Investigator, Zhaoping Li, Chief / Professor of Medicine, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 20-000879
Record Dates: First submitted 2020-05-13; First posted 2020-06-11 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: PreDiabetes
Keywords: glucose control; microbiome; prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: This is a double blinded, pilot placebo-controlled trial of two interventions compared to placebo to determine the effects individually of Metabolic Rheostat™ and Butyrate Ultra daily consumption for 8 weeks on glucose homeostasis in subjects with prediabetes. The study will include 20 subjects with prediabetes treated with Metabolic Rheostat™; 20 subjects with prediabetes treated with Butyrate Ultra and 20 subjects with prediabetes treated with placebo. Participants will take 6 capsules daily, two capsules three times per day 30 minutes prior to each meal for 56 days.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Metabolic Rheostat™ (Experimental): Participants will take 6 capsules of Rheostat daily, two capsules three times per day 30 minutes prior to each meal for 56 days.
  Interventions: Dietary Supplement: Metabolic Rheostat
- Butyrate Ultra (Experimental): Participants will take 6 capsules Butyrate Ultra daily, two capsules three times per day 30 minutes prior to each meal for 56 days.
  Interventions: Dietary Supplement: Butyrate Ultra
- Placebo (Placebo Comparator): Participants will take 6 capsules of placebo daily, two capsules three times per day 30 minutes prior to each meal for 56 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Metabolic Rheostat — Metabolic Rheostat™ Ingredients: Ginseng extract, Ginseng root extract, berberine chloride, Livaux (gold kiwi powder), MegaSporeBiotic, and MenaquinGold (vitamin K2-7) powder
  Arms: Metabolic Rheostat™
Dietary Supplement: Butyrate Ultra — An anerobic probiotic supplement that contains butyrate-producing Butyricicoccus pullicaecorum 25-3T, vitamin K2, and fenugreek to maintain healthy glucose balance.
  Arms: Butyrate Ultra
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to examine the effect of Metabolic Rheostat™ and Butyrate Ultra on blood glucose levels after a liquid meal challenge in patients with prediabetes. In addition, the study also aims to look at the effect of Metabolic Rheostat™ and Butyrate Ultra on weight, HgbA1c, fasting glucose, cholesterol, triglycerides, inflammation markers, and hormones.

DETAILED DESCRIPTION:
This is a double blinded, pilot placebo-controlled trial of two interventions compared to placebo to determine the effects individually of Metabolic Rheostat™ and Butyrate Ultra daily consumption for 8 weeks on glucose homeostasis in subjects with prediabetes. The entire study will last 10 weeks including screen. The study will include 20 subjects with prediabetes treated with Metabolic Rheostat™; 20 subjects with prediabetes treated with Butyrate Ultra and 20 subjects with prediabetes treated with placebo. Participants will take 6 capsules daily, two capsules three times per day 30 minutes prior to each meal for 56 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects with pre-diabetes.
2. Age> 18 years
3. Ability to understand and the willingness to sign a written informed consent.
4. Willing and able to comply with trial protocol and follow-up.

Exclusion Criteria:

1. Current use of any other investigational agent.
2. Current use of any agent for treatment of diabetes.
3. History of adverse effects, intolerance, or allergic reactions attributed to any medications.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Abnormal blood analysis for complete blood count (CBC), hepatic and renal injury tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Blood glucose effects of dietary supplement: Metabolic Rheostat vs. Butyrate Ultra | 2 hours
  Determine the effect of Metabolic Rheostat™ and Butyrate Ultra on blood glucose levels after a liquid meal challenge in patients with pre-diabetes.

SECONDARY OUTCOMES:
Metabolic impact of Metabolic Rheostat and Butyrate Ultra | 8 weeks
  Determining the effects of Metabolic Rheostat™ and Butyrate Ultra on gut hormones/incretins (including insulin, C-peptide, glucagon, CCK, GLP-1, GIP, and PYY) using Luminex bead-based technology.
Impact of Metabolic Rheostat and Butyrate Ultra on food addiction and cravings | 8 weeks
  Exploratory of Food Addiction (FA) using the Yale Food Addiction Scale (0 symptoms to 11 symptoms). Scale indications are: mild = 2-3 symptoms plus impairment or distress, moderate = 4-5 symptoms plus impairment or distress, severe = 6 or more symptoms plus impairment or distress).

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Center for Human Nutrition, 1000 Veteran Ave., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided